CLINICAL TRIAL: NCT03071159
Title: A Medium-term Evaluation of the Use, the Identified Problems, the Usability and the Effect on the Metabolic Control of the FreeStyle Flash Libre Glucose Monitoring System
Brief Title: An Evaluation of the FreeStyle Libre Flash Glucose Monitoring System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: JessaH
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-02

CONDITIONS: Flash Glucose Monitoring; Metabolic Control
Keywords: Flash Glucose Monitoring; Usability; Metabolic control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cases (Other): children (4-18 years) with type 1 diabetes mellitis using the FreeStyle Flash Libre glucose monitoring system (standard care)
  Interventions: Device: FreeStyle Flash Libre glucose monitoring system

INTERVENTIONS:
Device: FreeStyle Flash Libre glucose monitoring system — glucose monitoring system with sensors

SUMMARY:
Medium-term (6-12 months) evaluation of the use, the identified problems, the usability and the effect on the metabolic control of the FreeStyle Flash Libre glucose monitoring system in 90 children by questionnaires and routine measurement of HbA1c values.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitis
* Being followed in the Pediatric Diabetes Unit of the Jessa Hospital

Exclusion Criteria:

-

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-03-10 (Estimated); Study Completion 2018-03-10 (Estimated)

PRIMARY OUTCOMES:
Usability of the FreeStyle Flash Libre glucose monitoring system | 6-12 months follow up
  Usability of the FreeStyle Flash Libre glucose monitoring system by a questionnaire

SECONDARY OUTCOMES:
Problems associated with the FreeStyle Flash Libre glucose monitoring system | 6-12 months follow up
  Problems associated with the FreeStyle Flash Libre glucose monitoring system by a questionnaire
The effect of the FreeStyle Flash Libre glucose monitoring system on the metabolic control in patients | 6-12 months follow up
  The effect of the FreeStyle Flash Libre glucose monitoring system on the metabolic control in patients by measurement of the HbA1c values

CONTACTS AND LOCATIONS:
Overall Officials: Guy Massa, MD, PhD, Study Director — Department of Pediatric Diabetology, Jessa Ziekenhuis, Stadsomvaart 11, B3500
Locations (1):
- Jessa Hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No